CLINICAL TRIAL: NCT07282626
Title: Effectiveness of Active Brain Construction Program in Community-Dwelling Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 202310063RINA
Record Dates: First submitted 2024-11-18; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-11

CONDITIONS: Community Dwelling; Elderly Adults; Lifestyle Risk Reduction
Keywords: Elderly; Community health; Lifestyle intervention; Behavior Change Technique; coaching
MeSH Terms: conditions — Risk Reduction Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ABC program with coaching (Experimental): ABC program with coaching techniques
  Interventions: Behavioral: Active comparator (ABC Program)
- ABC program (Active Comparator): ABC program without coaching techniques
  Interventions: Behavioral: ABC program with coaching
- others (Sham Comparator): other programs such as exercise or art program
  Interventions: Behavioral: ABC program with coaching

INTERVENTIONS:
Behavioral: ABC program with coaching — This program lasts 12 weeks and 2 hours per week and targets community-dwelling older adults aged 60 and above, conducted by a trained occupational therapist or other professionals. The program consists of exercise (muscle strength, aerobic exercise, balance, and cognicise), cognition (attention, memory, spatial concept, language, calculation ability, and cognitive flexibility), and lifestyle factors modification (topics about cognition, exercise, sleep, health and Mediterranean diet, leisure activities, lifestyle arrangement, medication usage, chronic-disease management, fall prevention, emotion, stress, communication, social resources, and closing). Homework was assigned to the participants every week. Based on motivation theory and behavior change techniques, this program adopts behavior change techniques.
  Arms: ABC program; others
Behavioral: Active comparator (ABC Program) — This program lasts 12 weeks and 2 hours per week and targets community-dwelling older adults aged 55 and above, conducted by a trained occupational therapist or other professionals. The program consists of exercise (muscle strength, aerobic exercise, balance, and cognicise), cognition (attention, memory, spatial concept, language, calculation ability, and cognitive flexibility), and lifestyle factors modification (topics about cognition, exercise, sleep, health and Mediterranean diet, leisure activities, lifestyle arrangement, medication usage, chronic-disease management, fall prevention, emotion, stress, communication, social resources, and closing). Homework was assigned to the participants every week. Compared to the experiment group, there is no coaching techniques involved.
  Arms: ABC program with coaching

SUMMARY:
The urgency of health promotion and dementia prevention is paramount. In 2019, the World Health Organization announced the "Risk reduction of cognitive decline and dementia," which reviewed evidence-based prevention aspects and deduced 12 preventative dimensions, all related to lifestyle adjustments. Several are also related to chronic disease management. Therefore, referencing the theoretical foundation of chronic disease management and lifestyle interventions, and through the use of coaching skills-including goal setting, action planning, problem-solving, etc.-as indicators of effective behavior change, a 12-week group intervention program is developed for the prevention and delay of disability and dementia. This program aims to promote healthy behaviors, lifestyle changes, and cognitive function effects.

This study aims to investigate whether the "Active Brain Construction Program (ABC Program)," led by trainers with coaching skills, can promote behavior participation in a dementia-preventive healthy lifestyle among community-dwelling elders, as well as enhance their health status and cognitive function. Furthermore, it compares the cognitive enhancement effects on community-dwelling elders between the coached and non-coached "Active Brain Construction Program (ABC Program)" against a control group.

This study is a quasi-experimental non-randomized controlled trial, arranging three groups (experimental group, active control group, and control group) for comparison: 1) the coached "Brain-Healthy Lifestyle Reformation Course" group, 2) the general "Brain-Healthy Lifestyle Reformation Course" group, and 3) the control group (e.g., physical fitness class, nutrition courses). The elders undergo assessments before and after the course, including the collection of basic data. The primary effectiveness indicators are: the Health-Promoting Lifestyle Profile-Taiwan Short Form (HELP-T-SF) and the Goal Achievement Scale (GAS), with GAS measuring the experimental and active control groups; the secondary indicators include: the questionnaire for the Prevention and Delay of Disability Care for the Elderly (program effectiveness evaluation), the ICOPE Function Self-Assessment Scale for the Elderly - Self-Rating version, and the WHO-5 Well-Being Index. Data analysis collected includes: descriptive statistics of demographic baseline data, paired t-test comparisons of pre- and post-test differences within groups, ANOVA for between-group differences and post-hoc comparisons, and qualitative observational records to aid interpretation during the intervention process.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 55 and older
* reside in the community
* independently care for themselves and go outside to attend activities.
* can read and write sentences, comprehend conversations, and communicate appropriately.

Exclusion Criteria:

Individuals diagnosed with neurological conditions

* dementia
* mild cognitive impairment
* stroke.

Ages: 55 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 75 (Actual)
Dates: Start 2023-11-09 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Health Enhancement Lifestyle Profile -Taiwanese Version -Short Form | Perioperative/Periprocedural
  The original version contains a total of 56 items, categorized into the following subscales: 1) Exercise, 2) Diet, 3) Productive or Social Activities, 4) Leisure, 5) Activities of Daily Living, 6) Stress Management and Spiritual Participation, and 7) Other Health Promotion and Risk Behaviors. The complete original Taiwanese version consists of 59 items using a 3-point scale, and the HELP-T-SF consisted of 20 items, demonstrating acceptable internal consistency (Cronbach's alpha = 0.781) and test-retest reliability (ICC = 0.782). All items significantly correlated with the total score (0.303 to 0.535) and with the original HELP-T (0.749). Criterion-related validity showed moderate correlations with well-being and quality of life. The short form also resulted in significant time savings, requiring only 15-20 minutes to complete.

SECONDARY OUTCOMES:
Outcome Measurement of Health-Promotion Program for Community-Dwelling Elderly | Perioperative/Periprocedural
  The questionnaire consists of 20 items encompassing five dimensions: cognition, muscle strength, functional living, nutritional oral health, and psychosocial aspects, with four items dedicated to each dimension. The overall reliability and validity are good, with internal consistency (Cronbach's α = 0.82) and test-retest reliability (ICC = 0.927). The questionnaire shows a moderate correlation with the Kihon Checklist and can significantly distinguish between healthy individuals and those with dementia.
Integrated care for older people (ICOPE) | Perioperative/Periprocedural
  The assessment includes a total of 8 items across six key dimensions: cognition, behavior, nutrition, hearing, vision, and depression. If any responses indicate abnormalities, functional issues can be detected early, allowing for timely interventions such as exercise and nutritional management.

CONTACTS AND LOCATIONS:
Locations (1):
- Communities, Kaohsiung City, Taiwan